CLINICAL TRIAL: NCT02348333
Title: Seven-day Repeated Dose Clinical Pharmacological Study of FYU-981 Administered to Healthy Male Adults (Phase I Study).
Brief Title: Repeated Dose Phase I Study of FYU-981
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FYU-981-002
Record Dates: First submitted 2015-01-18; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
MeSH Terms: interventions — dotinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FYU-981 (Active Comparator)
  Interventions: Drug: FYU-981, (Oral daily dosing for 7 days)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo, (Oral daily dosing for 7 days)

INTERVENTIONS:
Drug: FYU-981, (Oral daily dosing for 7 days) — Subjects randomized to the FYU-981 arm receive active drug, FYU-981.
  Arms: FYU-981
Drug: Placebo, (Oral daily dosing for 7 days) — Subjects randomized to the placebo arm receive placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of 7-day-repeated doses of FYU-981 administered orally to healthy male adults once daily. Participants are randomized to placebo (n=3) or FYU-981 (n=6) in each step. After follow-up examination in the step of lower dose, the next dose is administered.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy adult subjects
* Body mass index: >=18.5 and <25.0

Exclusion Criteria:

* Subjects with any disease or any history of diseases that might be unsuitable for participation in the clinical study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax: Maximum plasma concentration) | 1-, 4-, and 7-day
Pharmacokinetics (Cmin: Minimum plasma concentration) | 1-, 2-, 3-, 4-, 5-, 6- and 7-day
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 1-, 4-, and 7-day
Pharmacokinetics (T1/2: Elimination half-life of plasma concentration) | 1-, 4-, and 7-day
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 1-, 4-, and 7-day
Pharmacokinetics (Rauc: Accumulation ratio of AUC0-24) | 4-, and 7-day
Pharmacokinetics (kel: Elimination rate constant) | 1-, 4-, and 7-day
Pharmacokinetics (CLtot/F: Total clearance / Fraction of dose absorbed) | 1-, 4-, and 7-day
Pharmacokinetics (Ae: Amount of drug excreted in urine) | 9 days
Pharmacokinetics (fe: Fraction of dose excreted in urine) | 9 days

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Tokyo, Japan